CLINICAL TRIAL: NCT04930133
Title: Totality Outcome of Afatinib Sequential Treatment in Patients With EGFR Sensitizing Mutation-positive NSCLC in South Korea
Brief Title: Retrospective Multi-cohort Study of Frontline Afatinib Followed by 2nd Line Therapy Including Osimertinib, Chemotherapy or Other Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Jin Hyoung Kang, Division of Medical Oncology, Department of Internal Medicine, Seoul St. Mary's Hospital
Other Study IDs: TOAST
Record Dates: First submitted 2021-06-13; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: NSCLC
Keywords: T790; afatinib
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A: T790M+ patients sequentially treated with osimertinib in cohort A
  Interventions: Drug: Gilotrif
- Cohort B: T790M- patients treated with chemotherapy or other treatments in cohort B
  Interventions: Drug: Gilotrif
- Cohort C: patients with unknown mutation status in cohort C
  Interventions: Drug: Gilotrif
- Cohort D: Cohort D included patients who were still ongoing with afatinib.
  Interventions: Drug: Gilotrif

INTERVENTIONS:
Drug: Gilotrif — This is non-interventional, multi-center, multi-cohort study based on existing data from EGFR sensitizing mutation-positive NSCLC patients treated with afatinib as the first-line treatment. Enrolled patients will be categorized into four cohorts (cohort A, B, C and D) according to the type of second line treatment with biopsy results before start of second line treatment.

SUMMARY:
The T790M mutation is highly sensitive to osimertinib, which is approved in this setting following failure of gefitinib, erlotinib or afatinib. In contrast to first- and second-generation EGFR TKIs, no predominant resistance mechanism to first-line osimertinib has been clearly defined yet. The most common mechanisms of resistance were c-MET amplification only for 15% of patients and the emergence of the EGFR C797S mutation in 7%, while > 60% of patients were still with no identifiable mechanisms of resistance. As a result, targeted treatment options following first-line osimertinib failure remain limited. Thus, interest on sequential administration of EGFR TKIs in patients with EGFR mutation-positive NSCLC has been growing. So, here in this study, we intend to investigate treatment outcome (TOT) along with the several treatment options starting from the first line EGFR TKI treatment to various second line treatments including 3rd generation TKI and chemotherapy and others.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years
2. Stage IIIB/IIIC/IV/IVA/IVB NSCLC patients treated with first-line afatinib for EGFR sensitizing mutations (Del19, L858R, G719X, S768I, or L861Q etc.)
3. Afatinib treatment was started 13 month prior to data collection date to reduce premature censoring of patients. Data cutoff date will be determined before data entry starts.

Exclusion Criteria:

1. Patients who received drug(s) other than afatinib (Giotrif®) as the first-line treatment
2. Patients who received drug(s) other than 3rd-generation EGFR TKI osimertinib as the second-line in "Cohort A'

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-interventional, multi-center, multi-cohort
Sampling Method: Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Total TOT | Non-interventional study (NIS) based on the existing data from patients' medical records(2013-08-01 ~ 2029-04-30).
  the time on treatment (total TOT) of EGFR M+ NSCLC patients treated with afatinib in the first-line (TOT-1) followed by second line treatments(TOT-2) including osimertinib, chemotherapy and other treatments.

SECONDARY OUTCOMES:
objective response rate (ORR-1 & ORR-2's) | Non-interventional study (NIS) based on the existing data from patients' medical records(2013-08-01 ~ 2029-04-30).
overall survival time | Non-interventional study (NIS) based on the existing data from patients' medical records(2013-08-01 ~ 2029-04-30).

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hyoung Kang, Study Chair — Seoul St. Mary's Hospital, The Catholic University of Korea
Locations (1):
- Jin Hyoung Kang, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided